CLINICAL TRIAL: NCT01113138
Title: Pharmacokinetic Study of Mablet as Oral Supplement and Magnesium Sulfate as Infusion
Brief Title: Study of the Metabolism of Two Magnesium Supplements in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Gunnar Kjems APS (Industry); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 9727b
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Clearance; Half-life; Absorption fraction; Pharmacokinetics
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (No Intervention)
- Mablet (Active Comparator)
  Interventions: Dietary Supplement: Mablet (Magnesium-supplement)
- Magnesium sulfate (Active Comparator)
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Dietary Supplement: Mablet (Magnesium-supplement) — Mablet: Magnesium hydroxide/ -oxide (360 mg/tablet) 3 tablets as a single dose Produced by: Gunnar Kjems APS
  Other Names: Mablet
  Arms: Mablet
Drug: Magnesium Sulfate — Solution for a single bolus-infusion, containing 2 grams of magnesium sulfate.
  Other Names: Magnesiumsulfat 'SAD'
  Arms: Magnesium sulfate

SUMMARY:
The present study is part of a project titled 'Magnesium in asthma and chronic obstructive pulmonary disease'. The hypothesis of the main project is that daily magnesium supplement will benefit patients with asthma and chronic obstructive pulmonary disease.

The aim of this part of the project is to study the pharmacokinetics of the following two magnesium supplements:

* Mablet (dietary supplement)
* Magnesium Sulfate (solution for infusion)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.

Exclusion Criteria:

* Smokers,
* Using pharmaceuticals/supplements,
* Vegans/vegetarians,
* Major changes in eating habits within one week prior to study start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Two years
  Clearance, half-life & absorption fraction

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Professor, Principal Investigator — Dept. of Respiratory Medicine, Aarhus University Hospital
Locations (1):
- Research Dept. of Respiratory Medicine, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Schlingmann KP, Konrad M, Seyberth HW. Genetics of hereditary disorders of magnesium homeostasis. Pediatr Nephrol. 2004 Jan;19(1):13-25. doi: 10.1007/s00467-003-1293-z. Epub 2003 Nov 22. PMID 14634861
- [Background] Beasley R, Aldington S. Magnesium in the treatment of asthma. Curr Opin Allergy Clin Immunol. 2007 Feb;7(1):107-10. doi: 10.1097/ACI.0b013e328012ce4b. PMID 17218820
- [Background] Emelyanov A, Fedoseev G, Barnes PJ. Reduced intracellular magnesium concentrations in asthmatic patients. Eur Respir J. 1999 Jan;13(1):38-40. doi: 10.1183/09031936.99.13103899. PMID 10836320
- [Background] Dominguez LJ, Barbagallo M, Di Lorenzo G, Drago A, Scola S, Morici G, Caruso C. Bronchial reactivity and intracellular magnesium: a possible mechanism for the bronchodilating effects of magnesium in asthma. Clin Sci (Lond). 1998 Aug;95(2):137-42. PMID 9680494
- [Background] Alamoudi OS. Hypomagnesaemia in chronic, stable asthmatics: prevalence, correlation with severity and hospitalization. Eur Respir J. 2000 Sep;16(3):427-31. doi: 10.1034/j.1399-3003.2000.016003427.x. PMID 11028655
- [Background] Bede O, Suranyi A, Pinter K, Szlavik M, Gyurkovits K. Urinary magnesium excretion in asthmatic children receiving magnesium supplementation: a randomized, placebo-controlled, double-blind study. Magnes Res. 2003 Dec;16(4):262-70. PMID 14979636
- [Background] Aziz HS, Blamoun AI, Shubair MK, Ismail MM, DeBari VA, Khan MA. Serum magnesium levels and acute exacerbation of chronic obstructive pulmonary disease: a retrospective study. Ann Clin Lab Sci. 2005 Autumn;35(4):423-7. PMID 16254259
- [Background] Rowe BH, Camargo CA Jr. The role of magnesium sulfate in the acute and chronic management of asthma. Curr Opin Pulm Med. 2008 Jan;14(1):70-6. doi: 10.1097/MCP.0b013e3282f19867. PMID 18043278
- [Background] Nasulewicz A, Zimowska W, Bayle D, Dzimira S, Madej J, Rayssiguier Y, Opolski A, Mazur A. Changes in gene expression in the lungs of Mg-deficient mice are related to an inflammatory process. Magnes Res. 2004 Dec;17(4):259-63. PMID 15726901
- [Background] Gontijo-Amaral C, Ribeiro MA, Gontijo LS, Condino-Neto A, Ribeiro JD. Oral magnesium supplementation in asthmatic children: a double-blind randomized placebo-controlled trial. Eur J Clin Nutr. 2007 Jan;61(1):54-60. doi: 10.1038/sj.ejcn.1602475. Epub 2006 Jun 21. PMID 16788707
- [Background] Fogarty A, Lewis SA, Scrivener SL, Antoniak M, Pacey S, Pringle M, Britton J. Oral magnesium and vitamin C supplements in asthma: a parallel group randomized placebo-controlled trial. Clin Exp Allergy. 2003 Oct;33(10):1355-9. doi: 10.1046/j.1365-2222.2003.01777.x. PMID 14519140
- [Background] Hill J, Micklewright A, Lewis S, Britton J. Investigation of the effect of short-term change in dietary magnesium intake in asthma. Eur Respir J. 1997 Oct;10(10):2225-9. doi: 10.1183/09031936.97.10102225. PMID 9387944
- [Background] Abreu Gonzalez J, Hernandez Garcia C, Abreu Gonzalez P, Martin Garcia C, Jimenez A. [Effect of intravenous magnesium sulfate on chronic obstructive pulmonary disease exacerbations requiring hospitalization: a randomized placebo-controlled trial]. Arch Bronconeumol. 2006 Aug;42(8):384-7. doi: 10.1016/s1579-2129(06)60551-x. Spanish. PMID 16948990